CLINICAL TRIAL: NCT02560181
Title: Pilot Study of Whole Gland Salvage HDR Prostate Brachytherapy for Locally Recurrent Prostate Cancer
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sunnybrook Health Sciences Centre (Other)
Responsible Party: Principal Investigator, Dr. Hans Chung, Radiation Oncologist, Sunnybrook Health Sciences Centre
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: clinicaltrials_hchu_180-2014
Record Dates: First submitted 2015-09-17; First posted 2015-09-25 (Estimated); Last update posted 2024-11-27 (Actual); Status verified 2024-11

CONDITIONS: Prostate Cancer Recurrent
Keywords: recurrent prostate cancer, HDR whole gland salvage
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- HDR whole gland salvage treatment (Other): Locally recurrent prostate cancer Whole gland HDR brachytherapy administered Whole gland dose=10.5Gy x 2 fractions delivered one week apart GTV dose=13.5Gy x 2 fractions delivered one week apart
  Interventions: Radiation: HDR brachytherapy

INTERVENTIONS:
Radiation: HDR brachytherapy — Whole gland salvage

SUMMARY:
Radiation therapy is considered a standard treatment option for the management of localized prostate cancer. Among the 20-30% of patients who recur, there is no consensus on the optimal salvage therapy. Salvage options available for isolated local recurrence include; temporary or permanent implantation of radioactive seeds into the prostate, complete removal of the prostate gland, use of low temperatures to treat the disease (cryotherapy), and high frequency ultrasound to treat the disease. There are risks of complications associated with all these treatments, and there is presently no consensus as to which treatment is the best. The aim of this pilot study is to look at the feasibility and toxicities of whole gland salvage treatment of the prostate using temporary implantation of radioactive seeds into the prostate.

DETAILED DESCRIPTION:
Radiation therapy is considered a standard treatment option for the management of localized prostate cancer. Among the 20-30% of patients who recur, there is no consensus on the optimal salvage therapy. Salvage options available for isolated local recurrence include; temporary or permanent implantation of radioactive seeds into the prostate, complete removal of the prostate gland, use of low temperatures to treat the disease (cryotherapy), and high frequency ultrasound to treat the disease. There are risks of complications associated with all these treatments, and there is presently no consensus as to which treatment is the best. The aim of this pilot study is to look at the feasibility and toxicities of whole gland salvage treatment of the prostate using temporary implantation of radioactive seeds into the prostate. Reports of the efficacy and toxicities of whole gland salvage HDR brachytherapy for local recurrence after external beam radiation therapy are limited to single-institution studies with small sample sizes. Given that our institution has the highest volume of prostate brachytherapy cases in Ontario and that we receive a significant number of referrals from other cancer centres for brachytherapy, this study will aim to add to the literature and help guide salvage therapy practice within our institution.

ELIGIBILITY:
Inclusion Criteria:

* Biopsy confirmed locally recurrent prostate adenocarcinoma > 30mths after completion of XRT by stereotactic transperineal biopsy
* Staging T2-weighted, DWI- and DCE- MRI that demonstrates recurrence confined to prostate, and correlates with stereotactic transperineal biopsy
* Previous external beam radiotherapy for prostate cancer with standard/conventional fractionation (1.8-2.0 Gy per fraction), or moderate hypofractionation (2.4-3.4 Gy per fraction).
* Staging CT or MRI (abdomen and pelvis) and bone scan are negative for metastases
* IPSS < 15
* Baseline (post XRT) serum PSA < 10ng/mL
* Prostate volume as measured by TRUS < 50cc
* ECOG performance status 0-1

Exclusion Criteria:

* Disease adjacent to the urethra as visible on MRI
* Any of the following prior therapies; TURP, radionuclide prostate brachytherapy, prostatectomy or prostatic cryosurgery, HIFU, bilateral orchiectomy, chemotherapy for prostatic carcinoma
* Evidence of castrate resistance (defined as PSA > 3ng/mL while testosterone is < 1.7nmol/L) Patients could have been on combined androgen blockade with initial XRT but are excluded if this was started due to PSA progression

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2014-08; Primary Completion 2027-08-30 (Estimated); Study Completion 2027-08-30 (Estimated)

PRIMARY OUTCOMES:
Acute GI toxicities | 3 mths post brachytherapy
  Acute GI toxicities using NCI CTCAE v4.0
Acute GU toxicities | 3 moths post brachytherapy
  Acute GU toxicities utilizing NCI CTCAE v4.0

SECONDARY OUTCOMES:
Acute GU symptoms | 5 years
  Acute GU symptoms American Urological Association Symptom Index Score (IPSS)
Late GU symptoms | 5 years
  Late GU symptoms American Urological Association Symptom Index Score (IPSS)
Late GI toxicities | 5 years
  Late GI toxicities using NCI CTCAE v.4.0
Late GU toxicities | 5 years
  Late GU Toxicities using NCI CTCAE v.4.0
Biochemical disease free survival | 5 years
  PSA
Quality of Life (QoL) | 5 years
  QoL measured using Expanded Prostate Cancer Index Composite (EPIC)

CONTACTS AND LOCATIONS:
Overall Officials: Hans Chung, MD, Principal Investigator — Odette Cancer Centre, Sunnybrook Health Sciences Centre
Locations (1):
- Odette Cancer Centre, Sunnybrook Health Sciences Centre, Toronto, Ontario, Canada